CLINICAL TRIAL: NCT07071818
Title: Evaluation of the Vesicourethral Angle by Preoperative and Postoperative Transperineal Ultrasound in Patients Undergoing Colpocleisis Surgery and Assessment of de Novo Urinary Incontinence
Brief Title: Transperineal Ultrasound Evaluation of Vesicourethral Angle and de Novo SUI After Colpocleisis Surgery
Acronym: colpocleisis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Serkan Kumbasar, ASSOCIATE PROFESSOR, Gaziosmanpasa Research and Education Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: gopcolpoultra
Record Dates: First submitted 2025-07-04; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Prolapse, Vaginal
Keywords: Colpocleisis; Transperineal Ultrasound; de Novo Incontinence; Vesicourethral Angle
MeSH Terms: conditions — Uterine Prolapse

STUDY DESIGN:
Intervention Model Description: This is a prospective, observational cohort study designed to evaluate anatomical and functional changes in patients undergoing colpocleisis surgery. Patients will be followed at predefined intervals (preoperative, 1 month, and 6 months postoperatively) to assess changes in the vesicourethral angle using transperineal ultrasound, and to determine the incidence of de novo stress urinary incontinence. The same cohort of patients will be observed over time without any randomization or intervention beyond standard surgical care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Colpocleisis Group (Other): This study has a single intervention cohort consisting of patients undergoing colpocleisis. All participants in this group will receive standard surgical care (colpocleisis), and no additional intervention will be administered as part of the research. The same protocol will be applied to all participants: vesicourethral angle will be measured using transperineal ultrasound before and six months after surgery. There is no comparison group or randomization.
  Interventions: Procedure: Colpocleisis Group

INTERVENTIONS:
Procedure: Colpocleisis Group — Participants will undergo colpocleisis surgery as part of routine clinical care. The study involves transperineal ultrasound (TPUS) to measure the vesicourethral angle preoperatively and postoperatively, along with assessments for de novo stress urinary incontinence, POP-Q staging, PFDI-20 questionnaire, and stress testing.

SUMMARY:
This prospective observational study aims to evaluate changes in the vesicourethral angle using transperineal ultrasound before and after colpocleisis surgery, and to assess the relationship of these changes with the development of de novo stress urinary incontinence.

DETAILED DESCRIPTION:
Colpocleisis is a surgical method used for treating pelvic organ prolapse (POP) in elderly women who are no longer sexually active. POP may mask stress urinary incontinence (SUI) by affecting urethral support. After colpocleisis, correction of the prolapse may alter the vesicourethral angle, potentially leading to de novo urinary incontinence.

This prospective observational study aims to evaluate changes in the vesicourethral angle using transperineal ultrasound (TPUS) before and after colpocleisis surgery, and to investigate its association with new-onset urinary incontinence. Assessments will be conducted at three time points: Preoperative Visit: Clinical evaluation, POP-Q measurements, PFDI-20 questionnaire, stress test, and TPUS measurement of the vesicourethral angle.

Postoperative 1st Month: General recovery and healing assessment. Postoperative 6th Month: Repeat POP-Q, PFDI-20, stress test, TPUS, and evaluation for de novo SUI.

The study aims to explore the role of TPUS in identifying anatomical changes that may contribute to urinary symptoms following colpocleisis.

ELIGIBILITY:
Inclusion Criteria:

Postmenopausal women with stage 3 or 4 pelvic organ prolapse (according to POP-Q score), who are not sexually active and do not desire future vaginal intercourse, and who consent to undergo colpocleisis surgery will be included in the study.

Exclusion Criteria:

Those with a history of stress incontinence surgery Those who underwent an additional vesicourethral intervention in addition to colpocleisis surgery Those who wanted sexual intercourse

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Vesicourethral Angle Measured by Transperineal Ultrasound | Baseline (Preoperative), 6 Months Postoperative
  The primary outcome is the change in the vesicourethral angle measured via transperineal ultrasound before and after colpocleisis surgery. The angle will be measured in degrees using standardized TPUS imaging protocols.
Incidence of de Novo Stress Urinary Incontinence | 6 Months Postoperative
  The proportion of patients who develop new-onset (de novo) stress urinary incontinence following colpocleisis surgery, as determined by physical examination (stress test) and patient-reported symptoms.
Change in PFDI-20 (Pelvic Floor Distress Inventory-20) Score | Preoperative, 6 Months Postoperative
  Evaluation of changes in pelvic floor symptoms and distress based on patient responses to the validated PFDI-20 questionnaire administered before and after surgery.
Change in POP-Q Stage | Preoperative, 6 Months Postoperative
  Assessment of anatomical improvement in pelvic organ prolapse using POP-Q staging system, comparing pre- and postoperative values.

CONTACTS AND LOCATIONS:
Overall Officials: ecenur çelikoğlu, md, Principal Investigator — Gaziosmanpaşa training and research hospital; yağmur acıyiyen, md, Principal Investigator — Gaziosmanpaşa training and research hospital
Locations (1):
- Gaziosmanpaşa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No